CLINICAL TRIAL: NCT01218958
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Medisorb® Naltrexone in Alcohol-Dependent Adults
Brief Title: ALK21-003: Study of Medisorb® Naltrexone (VIVITROL®) in Alcohol-Dependent Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Bernard Silverman, MD, Vice President, Clinical Development, Alkermes, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK21-003
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Results first posted 2010-12-07 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Alcoholism
Keywords: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; vivitrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Medisorb naltrexone 190 mg (Experimental)
  Interventions: Drug: Medisorb naltrexone 190 mg
- Medisorb naltrexone 380 mg (Experimental)
  Interventions: Drug: Medisorb naltrexone 380 mg
- Placebo for Medisorb naltrexone 190 mg (Placebo Comparator)
  Interventions: Drug: Placebo matching Medisorb naltrexone 190 mg
- Placebo for Medisorb naltrexone 380 mg (Placebo Comparator)
  Interventions: Drug: Placebo matching Medisorb naltrexone 380 mg

INTERVENTIONS:
Drug: Medisorb naltrexone 190 mg — Intramuscular (IM) injection once every 4 weeks for a total of 6 administrations.
  Other Names: naltrexone for extended-release injectable suspension
  Arms: Medisorb naltrexone 190 mg
Drug: Medisorb naltrexone 380 mg — IM injection once every 4 weeks for a total of 6 administrations.
  Other Names: VIVITROL 380 mg; naltrexone for extended-release injectable suspension
  Arms: Medisorb naltrexone 380 mg
Drug: Placebo matching Medisorb naltrexone 190 mg — IM injection once every 4 weeks for a total of 6 administrations.
  Arms: Placebo for Medisorb naltrexone 190 mg
Drug: Placebo matching Medisorb naltrexone 380 mg — IM injection once every 4 weeks for a total of 6 administrations.
  Other Names: Placebo matching VIVITROL 380 mg
  Arms: Placebo for Medisorb naltrexone 380 mg

SUMMARY:
This was a Phase 3, multicenter, randomized, double-blind, placebo-controlled study conducted in subjects diagnosed with alcohol dependence as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Ed. (DSM-IV). Subjects were randomized (2:2:1:1) to receive intramuscular (IM) injections of Medisorb® naltrexone 190 mg, Medisorb naltrexone 380 mg, placebo for Medisorb naltrexone 190 mg, or placebo for Medisorb naltrexone 380 mg (VIVITROL®). Study drug was administered every 4 weeks for a total of 6 injections.

DETAILED DESCRIPTION:
All subjects received standardized biopsychosocial support therapy (BRENDA Approach [Volpicelli, JR [2001]; Guilford Press: New York]) at each visit.

Subjects who completed this study (ie, received 6 injections of study drug and completed all study visits) and continued to meet eligibility criteria were given the option to enroll in extension study ALK21-003EXT (NCT01218971). A second extension, Study ALK21-010 (NCT00156923), was conducted subsequent to ALK21-003EXT.

ELIGIBILITY:
Primary Inclusion Criteria:

* Diagnosis of alcohol dependence based on Diagnostic and Statistical Manual of Mental Disorders, 4th Ed. (DSM-IV) criteria
* Male or non-pregnant, non-lactating female
* Able to provide TimeLine Follow-Back (TLFB) alcohol consumption information for 90-day period before detoxification and/or screening
* At least 2 episodes of heavy alcohol drinking per week during the 30 days before detoxification and/or screening
* Negative urine toxicological screen for opiates on day of randomization
* Noncustodial, stable residence and phone plus 1 contact with verifiable address and phone

Primary Exclusion Criteria:

* Evidence of hepatic failure including: ascites, prolonged prothrombin time (PT) (international normalized ratio [INR] ≥1.7), bilirubin >10% above upper limit of normal (ULN) and/or esophageal variceal disease
* Active hepatitis and/or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) higher than 3xULN
* History of pancreatitis
* Major depression with suicidal ideation, psychosis, bipolar disorder, or psychiatric disorders that would compromise subject's ability to complete the study
* Current dependence (within past year) per DSM-IV criteria to benzodiazepines, opioids or cocaine
* Use of benzodiazepines and/or Ambien® (zolpidem tartrate) within 7 days prior to first dose of study medication
* Greater than 7 days inpatient treatment for substance use disorders within 30 days of randomization
* Use of any opioids and/or methadone within 14 days of screening, or likely requiring opioid therapy during study period
* Use of oral naltrexone or disulfiram within 14 days of screening
* Known intolerance and/or hypersensitivity to naltrexone, carboxymethylcellulose, or polylactide-co-glycolide (PLG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2002-02; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Silverman, MD, Study Director — Alkermes, Inc.

REFERENCES:
- [Result] Garbutt JC, Kranzler HR, O'Malley SS, Gastfriend DR, Pettinati HM, Silverman BL, Loewy JW, Ehrich EW; Vivitrex Study Group. Efficacy and tolerability of long-acting injectable naltrexone for alcohol dependence: a randomized controlled trial. JAMA. 2005 Apr 6;293(13):1617-25. doi: 10.1001/jama.293.13.1617. PMID 15811981
- [Result] O'Malley SS, Garbutt JC, Gastfriend DR, Dong Q, Kranzler HR. Efficacy of extended-release naltrexone in alcohol-dependent patients who are abstinent before treatment. J Clin Psychopharmacol. 2007 Oct;27(5):507-12. doi: 10.1097/jcp.0b013e31814ce50d. PMID 17873686
- [Result] Gastfriend DR, Garbutt JC, Pettinati HM, Forman RF. Reduction in heavy drinking as a treatment outcome in alcohol dependence. J Subst Abuse Treat. 2007 Jul;33(1):71-80. doi: 10.1016/j.jsat.2006.09.008. Epub 2007 Feb 22. PMID 17588491
- [Result] Lucey MR, Silverman BL, Illeperuma A, O'Brien CP. Hepatic safety of once-monthly injectable extended-release naltrexone administered to actively drinking alcoholics. Alcohol Clin Exp Res. 2008 Mar;32(3):498-504. doi: 10.1111/j.1530-0277.2007.00593.x. Epub 2008 Jan 30. PMID 18241321
- [Result] Ciraulo DA, Dong Q, Silverman BL, Gastfriend DR, Pettinati HM. Early treatment response in alcohol dependence with extended-release naltrexone. J Clin Psychiatry. 2008 Feb;69(2):190-5. doi: 10.4088/jcp.v69n0204. PMID 18348601
- [Result] Pettinati HM, Gastfriend DR, Dong Q, Kranzler HR, O'Malley SS. Effect of extended-release naltrexone (XR-NTX) on quality of life in alcohol-dependent patients. Alcohol Clin Exp Res. 2009 Feb;33(2):350-6. doi: 10.1111/j.1530-0277.2008.00843.x. Epub 2008 Nov 25. PMID 19053979
- [Result] Lapham S, Forman R, Alexander M, Illeperuma A, Bohn MJ. The effects of extended-release naltrexone on holiday drinking in alcohol-dependent patients. J Subst Abuse Treat. 2009 Jan;36(1):1-6. doi: 10.1016/j.jsat.2008.07.001. Epub 2008 Sep 4. PMID 18775624
- [Result] Cisler RA, Silverman BL, Gromov I, Gastfriend DR. Impact of treatment with intramuscular, injectable, extended-release naltrexone on counseling and support group participation in patients with alcohol dependence. J Addict Med. 2010 Sep;4(3):181-5. doi: 10.1097/ADM.0b013e3181c82207. PMID 21769033
- [Result] Pettinati HM, Silverman BL, Battisti JJ, Forman R, Schweizer E, Gastfriend DR. Efficacy of extended-release naltrexone in patients with relatively higher severity of alcohol dependence. Alcohol Clin Exp Res. 2011 Oct;35(10):1804-11. doi: 10.1111/j.1530-0277.2011.01524.x. Epub 2011 May 16. PMID 21575016

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects were screened up to 14 days before administration of study drug (Study Day 0).
Pre-assignment Details: A dynamic randomization was implemented to optimize balancing treatment assignment for 4 prespecified factors: gender, subject's baseline goal of abstinence (ie, yes/no), presence of abstinence prior to randomization, and study site.
Groups:
- Placebo Groups (Pooled): Results for the two groups that received placebo were pooled together for reporting purposes.
Period: Overall Study
Arm/Group | Medisorb Naltrexone 190 mg | Medisorb Naltrexone 380 mg | Placebo Groups (Pooled)
Started | 210 | 205 | 209
Completed | 126 | 124 | 128
Not Completed | 84 | 81 | 81

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medisorb Naltrexone 190 mg | Medisorb Naltrexone 380 mg | Placebo Groups (Pooled) | Total
Number analyzed (Participants) | 210 | 205 | 209 | 624
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 203 | 200 | 199 | 602
  >=65 years | 7 | 5 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (10.8) | 45.0 (10.1) | 44.7 (10.8) | 44.7 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 67 | 66 | 201
  Male | 142 | 138 | 143 | 423
Region of Enrollment [Number; unit: participants]
  United States | 210 | 205 | 209 | 624

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Heavy Drinking Days Over the Treatment Period
Description: Drinking rates were assessed from participants' self-reports using the validated Timeline Follow-Back (TLFB) method. Using a TLFB calendar, participants reported the number of days they had consumed alcohol along with the amount they consumed on each day. A heavy drinking day was defined as ≥5 drinks/day for men and ≥4 drinks/day for women.
Time Frame: Baseline through Week 24 (168 days)
Population: The last post-baseline observation carried forward (LOCF) of each participant in the intent-to-treat population (all randomized participants who received at least 1 injection of study drug) were utilized for the primary efficacy analysis.
Measure: Median (Inter-Quartile Range); unit: Percentage of days
Units Other Than Participants: Days
Arm/Group | Medisorb Naltrexone 190 mg | Medisorb Naltrexone 380 mg | Placebo Groups (Pooled)
Number analyzed (Participants) | 206 | 201 | 204
Number analyzed (Days) | 168 | 168 | 168
Percentage of days | 14.75 [3.23 to 44.58] | 10.23 [1.16 to 33.33] | 19.77 [6.01 to 50.15]
Statistical Analysis 1: Comparison: Medisorb Naltrexone 380 mg vs Placebo Groups (Pooled); The event rate (percentage) is represented by the number of heavy drinking days divided by number of days at risk. For each day, the active groups' results were contrasted with placebo to form the event rate ratio. Thus, a hazard ratio of 0.75 for the 380 mg group indicates a 25% reduction in heavy drinking compared with that of placebo. The method of analysis estimates the average ratio over time and accounts for discontinuation. Point/interval estimates for pairwise ratios were derived; Test type: Superiority or Other; p = 0.0245, Andersen-Gill recurrent-event Cox — The Hochberg method was used to adjust P-value for multiple comparisons (ie, 380 mg dose vs. placebo and 190 mg dose vs. placebo); Hazard Ratio (HR) = 0.751, 95% CI 2-sided [0.600 to 0.940]
Statistical Analysis 2: Comparison: Medisorb Naltrexone 190 mg vs Placebo Groups (Pooled); Test type: Superiority or Other; p = 0.0744, Andersen-Gill recurrent-event Cox model; Hazard Ratio (HR) = 0.830, 95% CI 2-sided [0.677 to 1.018]

2. Secondary Outcome: Number of Participants Reporting at Least 1 Treatment-emergent Adverse Event (TEAE)
Description: A TEAE is any adverse event, whether or not considered drug-related, that develops or worsens in severity after study drug administration begins (ie, from the first administration through the end of the follow-up period).
Time Frame: 24 weeks (Baseline to Week 24)
Measure: Number; unit: Participants
Arm/Group | Medisorb Naltrexone 190 mg | Medisorb Naltrexone 380 mg | Placebo Groups (Pooled)
Number analyzed (Participants) | 210 | 205 | 209
Participants | 190 | 187 | 181

ADVERSE EVENTS:
Time Frame: Events were recorded starting at baseline through 42 days after the last dose of study drug.
Arm/Group | Medisorb Naltrexone 190 mg | Medisorb Naltrexone 380 mg | Placebo Groups (Pooled)
Serious Adverse Events (participants affected / at risk) | 10/210 | 11/205 | 15/209
Other Adverse Events (participants affected / at risk) | 190/210 | 187/205 | 181/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medisorb Naltrexone 190 mg (N=210) | Medisorb Naltrexone 380 mg (N=205) | Placebo Groups (Pooled) (N=209)
Alcoholism (Psychiatric disorders) | 5 | 4 | 7
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0
Emotional distress (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder NOS (Psychiatric disorders) | 0 | 0 | 1
Pneumonia NOS (Infections and infestations) | 1 | 0 | 1
Interstitial pneumonia (Infections and infestations) | 0 | 1 | 0
Atrial fibrillation aggravated (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage NOS (Gastrointestinal disorders) | 0 | 1 | 0
Perirectal abscess (Gastrointestinal disorders) | 0 | 1 | 0
Chest tightness (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Inflammatory carcinoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Laryngeal cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Intervertebral disc herniation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Eosinophilic pneumonia acute (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Medisorb Naltrexone 190 mg (N=210) | Medisorb Naltrexone 380 mg (N=205) | Placebo Groups (Pooled) (N=209)
Nausea (Gastrointestinal disorders) | 53 | 68 | 23
Diarrhoea NOS (Gastrointestinal disorders) | 23 | 26 | 18
Vomiting NOS (Gastrointestinal disorders) | 22 | 28 | 12
Abdominal pain upper (Gastrointestinal disorders) | 17 | 8 | 9
Abdominal pain NOS (Gastrointestinal disorders) | 5 | 13 | 3
Dyspepsia (Gastrointestinal disorders) | 5 | 3 | 11
Injection site pain (General disorders) | 19 | 24 | 12
Fatigue (General disorders) | 34 | 41 | 23
Injection site induration (General disorders) | 7 | 13 | 4
Nasopharyngitis (Infections and infestations) | 32 | 22 | 23
Upper respiratory tract infection NOS (Infections and infestations) | 15 | 21 | 18
Insomnia (Psychiatric disorders) | 27 | 28 | 25
Anxiety NEC (Psychiatric disorders) | 10 | 13 | 12
Depression (Psychiatric disorders) | 3 | 16 | 8
Libido decreased (Psychiatric disorders) | 3 | 11 | 2
Headache NOS (Nervous system disorders) | 33 | 45 | 34
Dizziness (Nervous system disorders) | 23 | 26 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 19 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 9 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 8 | 11
Pain in limb (Musculoskeletal and connective tissue disorders) | 2 | 13 | 6
Appetite decreased NOS (Metabolism and nutrition disorders) | 12 | 26 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should a PI wish to disclose results, the Sponsor will review the results communications prior to public release and can embargo results communications for a period of at least 30 days prior to the submission, for review and approval. Revisions will be negotiated in good faith by the Investigator and Sponsor and may be submitted for publication or disclosed by the Investigator only following receipt of written approval from the Sponsor.